CLINICAL TRIAL: NCT04193891
Title: The Effect of Ketogenic Dietary Therapy on Sleep in Adult Epilepsy: a Pilot Study.
Brief Title: The Effect of Ketogenic Dietary Therapy on Sleep in Adult Epilepsy
Status: Terminated | Type: Observational
Why Stopped: due to COVID-19
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Institute for Clinical and Translational Research (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-1033; A535100 (Other: UW Madison); SMPH/NEUROLOGY/NEUROLOGY (Other: UW Madison); 5UL1TR002373-03 (NIH); Protocol Version 3/8/2020 (Other: UW Madison)
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; Seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Diet Group: Participants choosing to newly initiate the modified Atkins diet, a high fat low carb diet, for improved epilepsy control.
  Interventions: Other: Modified Atkins Diet
- Control Group: Participants not choosing to initiate dietary therapy for epilepsy. The participants in the control group will continue with the treatment regimen they have chosen together with their physician.

INTERVENTIONS:
Other: Modified Atkins Diet — The ketogenic diet, where individuals restrict their carbohydrate intake and significantly increase their intake of fats, was initially primarily used in children with severe epilepsy, often due to genetic syndromes. Recently, with the advent of slightly less restrictive forms of ketogenic dietary therapy (e.g. the modified Atkins diet), it has begun to be used in adults with intractable seizures who are not surgical candidates.
  Groups: Diet Group

SUMMARY:
The modified Atkins diet, a form of ketogenic therapy in which individuals severely restrict their carbohydrate intake and subsequently enter ketosis, has begun to be used as an adjunctive treatment in adults with intractable epilepsy who are not surgical candidates. In this study, the investigators examine the effect of ketogenic dietary therapy on sleep, as sleep deprivation is one of the most common seizure triggers and seizures themselves have been found to affect sleep quality. This pilot study will enroll twenty participants, ten of whom are initiating ketogenic dietary therapy and ten participants who are being treated with standard anti-seizure drug therapy.

DETAILED DESCRIPTION:
Twenty participants, 10 participants on the modified Atkins diet and 10 control participants, will be enrolled in the study. All participants will fill out validated sleep questionnaires and complete sleep and seizure diaries. Furthermore, all participants will wear actigraphy watches prior to ketogenic dietary therapy initiation as well as four to six weeks after being on the diet. For control participants, the actigraphy will be completed at two time points to mimic that of the participants in the dietary therapy group. For the home sleep studies for the subset of participants, these will be completed at similar time intervals as that of the actigraphy. Adherence to the diet will be monitored according to standard medical management; for any participant on the diet, he or she will keep track of food intake and track ketones, which will be submitted at the four to six week follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy

  * Diet arm - participants who plan to newly initiate treatment with the Modified Atkins Diet (MAD) within the next 2 months as an adjunctive treatment for epilepsy
  * Control arm - participants who do not plan to initiate ketogenic dietary therapy in the next 6 months

Exclusion Criteria:

* Diagnosed sleep disorders (obstructive sleep apnea, primary insomnia, idiopathic hypersomnia, narcolepsy type I or II, REM sleep behavior disorder)
* Previously attempted dietary therapy for epilepsy who were not successful or compliant
* Anticipated need to adjust anti-seizure medications within the next 3 months
* Already on a ketogenic diet at the beginning of the study
* Planning to pursue surgical treatment for epilepsy in the next 6 months
* Non-English speakers
* Standard modified Atkins diet exclusion criteria (see below)
* At the discretion of the PI
* Live greater than 20 miles from the greater Madison area (in case there is a need to personally pick up the home sleep monitor at the participant's home)
* More than two no show appointments in the past 6 months

For reference, the clinical exclusion criteria for the modified Atkins diet are listed here. These will have been verified clinically in order for the participant to be on the diet, and any reassessment of these criteria will be solely standard care, for clinical purposes:

* Unwilling to restrict carbohydrates
* Significantly underweight (BMI <18.5)
* Kidney disease
* Metabolic or mitochondrial disorder
* Pregnancy
* Aversion to liquids or inability to eat solid food
* At the discretion of the PI

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients receiving care in the epilepsy clinics at the University of Wisconsin School of Medicine and Public Health.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Change in Epworth Sleepiness Scale | before entering the study, 4-6 weeks after being on the diet (or 4-6 weeks after enrollment for control subjects)
  The Epworth Sleepiness Scale is a survey where participants score their chance of dozing (0-3, where 0 is 'would never doze', 1 is 'slight chance of dozing', 2 is 'moderate chance of dozing', and 3 is 'high chance of dozing') in 8 different situations. The total range in scores is 0-24 where higher scores indicate higher chances of dozing.
Change in Pittsburgh Sleep Quality Index | before entering the study, 4-6 weeks after being on the diet (or 4-6 weeks after enrollment for control subjects)
  The Pittsburgh Sleep Quality Index measures participant quality of sleep in each of 7 domains over the last month: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The total possible range of scores is 0-21 with 0 indicating no difficulties and 21 indicating severe difficulties.
Change in Morning-Eveningness Questionnaire | before entering the study, 4-6 weeks after being on the diet (or 4-6 weeks after enrollment for control subjects)
  The Morning-Eveningness Questionnaire is a 19-item survey that measures participant tendency toward being a 'morning' or 'evening' person. The total possible range of scores is 16-86 with scores of 41 and below indicating 'evening' types, scores between 42-58 being 'intermediate' types, and scores of 59 and above 'morning' types.
Change in Mean Sleep Time Per Night | before entering the study, 4-6 weeks after being on the diet (or 4-6 weeks after enrollment for control subjects)
  Measured via Fitbit and per participant sleep log report between four nights at baseline and four nights at follow-up
Change in Sleep Change Composition | before entering the study, 4-6 weeks after being on the diet (or 4-6 weeks after enrollment for control subjects)
  Using the Prodigy sleep system (Cerebra Health Inc.), which uses EEG, Electromyography (EMG), and Electrooculogram (EOG) to measure sleep, we will determine the amount of time spent in the various stages of sleep (REM, Non-Rapid Eye Movement (NREM) Stage 1, NREM Stage 2, NREM Stage 3)
Change in Sleep Latency | before entering the study, 4-6 weeks after being on the diet (or 4-6 weeks after enrollment for control subjects)
  Sleep latency is the time it takes to fall asleep. This will be measured using the Prodigy sleep system (Cerebra Health Inc.) using EEG, EMG, and EOG
Change in Number of Awakenings per Night | before entering the study, 4-6 weeks after being on the diet (or 4-6 weeks after enrollment for control subjects)
  This is the amount of times a participant is recorded as awake via the Prodigy (Cerebra Health Inc.) sleep system, according to EEG, EMG and EOG.
Change in Sleep Depth | before entering the study, 4-6 weeks after being on the diet (or 4-6 weeks after enrollment for control subjects)
  Sleep depth is a metric developed and patented by the company that is the maker of the Prodigy sleep system (Cerebra Health Inc.). It is a metric that estimates the ratio of time spent in light and deep sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Felton, MD/PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Felton EA, Cervenka MC. Dietary therapy is the best option for refractory nonsurgical epilepsy. Epilepsia. 2015 Sep;56(9):1325-9. doi: 10.1111/epi.13075. Epub 2015 Jul 22. PMID 26198999